CLINICAL TRIAL: NCT04037722
Title: Echocardiographic Changes After Oral Intake of 3-hydroxy Butyrate+Whey in a Human Endotoxemia Model
Brief Title: Echocardiographic Changes After 3-hydroxy Butyrate+Whey Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Arla Food Ingredients, Arla Viby. (Unknown); Aarhus University Hospital Skejby (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Ketone Heart Study
Record Dates: First submitted 2019-07-11; First posted 2019-07-30 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2019-07

CONDITIONS: Cardiac Output; Endotoxemia; Catabolic State; Echocardiography
Keywords: Cardiac Output; Endotoxemia; Ketone bodies; 3-hydroxy butyrate; Whey protein; Catabolic State
MeSH Terms: conditions — Endotoxemia | interventions — Whey

STUDY DESIGN:
Intervention Model Description: In a randomized crossover design, eight healthy lean young men will undergo either:
  i) Healthy conditions (overnight fast) + whey protein
  ii) Catabolic conditions (Inflammation (LPS) + 36-hour fast and bed rest) + whey protein
  iii) Catabolic conditions (Inflammation (LPS) + 36-hour fast and bed rest) + 3-OHB/whey protein
Who Masked: Participant, Outcomes Assessor
Masking Description: Interventions (saline/LPS) or whey/3-OHB+whey will be given by the investigator, and the echocardiography will be performed by another blinded investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy + Whey (Experimental): Healthy conditions (overnight fast)
  Interventions: Dietary Supplement: Whey
- Catabolic + Whey (Experimental): Catabolic conditions (36-hour fast, bed rest and inflammation (LPS))
  Interventions: Dietary Supplement: Whey
- Catabolic + 3-OHB / Whey (Experimental): Catabolic conditions (36-hour fast, bed rest and inflammation (LPS))
  Interventions: Dietary Supplement: 3-OHB + Whey

INTERVENTIONS:
Dietary Supplement: Whey — 45 g whey + 20 g maltodextrin
  Arms: Catabolic + Whey; Healthy + Whey
Dietary Supplement: 3-OHB + Whey — 50 g ketone + 45 g whey + 20 g maltodextrin
  Arms: Catabolic + 3-OHB / Whey

SUMMARY:
This study evaluates the cardiovascular effects of adding the ketone body 3-hydroxy butyrate (3-OHB) to whey protein during human endotoxemia. Further, this study compares cardiovascular changes during healthy and catabolic conditions.

Participants will receive isocaloric, isonitrogenous beverages of either whey or 3-OHB+whey in a randomized crossover design during either healthy (overnight fast) or catabolic conditions (inflammation/endotoxemia + 36 h fast and bed rest).

DETAILED DESCRIPTION:
Background: A newly published study found beneficial cardiovascular effects of 3-OHB infusion in a population with chronic heart failure, significantly increasing cardiac output. Similar effects on cardiac output were observed in healthy volunteers. These findings pave the way for 3-OHB as a therapeutic nutritional supplement, since it is well-absorbed during oral consumption. However, it is unknown whether the cardiovascular effects of 3-OHB persist during a sepsis-like catabolic state and when administered orally.

Aim: This study aims to investigate the cardiovascular effects of adding the ketone body 3-hydroxy butyrate (3-OHB) to whey protein during a human disease model, comprising endotoxemia + bed rest + fast.

Hypothesis:

1. Adding the ketone body 3-OHB to an oral protein supplement increases cardiac output measures
2. Catabolic stress (endotoxemia/inflammation + 36 h fast and bed rest) induces cardiovascular changes compared with healthy conditions (overnight fast)

   Interventions:

   In a randomized crossover design, eight healthy, lean, young men will undergo either:

   i) Healthy conditions (overnight fast) + whey protein^

   ii) Catabolic conditions (Inflammation (LPS) + 36-hour fast and bed rest*) + whey protein^

   iii) Catabolic conditions (Inflammation (LPS) + 36-hour fast and bed rest*) + 3-OHB/whey protein^"

   *LPS will be administered (1 ng/kg) the day prior to the study together with fast and bed rest. On the study day LPS (0.5 ng/kg) will be injected.

   ^Beverages will be isonitrogenous and isocaloric (fat will be added) with 45 g whey protein + 20 g maltodextrin. Bolus/sip administration will be applied (1/3 bolus, 1/2 sip)

   " 50 grams of 3-OHB will be orally administered (1/2 bolus, 1/2 sip)

ELIGIBILITY:
Inclusion Criteria:

* Between 20-40 years of age
* Body mass index between 20-30 kg/m^2
* Healthy
* Oral and written consent forms obtained prior to study day

Exclusion Criteria:

* Recent immobilization of an extremity that is not fully rehabilitated
* Lactose, lidocain or rubber allergies
* Current disease
* Use of anabolic steroids
* Smoking
* Former major abdominal surgery (Or current problems with the GI tract)

  •>10 hours of exercise/weak
* Present ketogenic diets or high-protein diets
* Blood doner that does not want to discontinue blood donations until study completion
* Pending MR scan

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-01-23 (Actual)

PRIMARY OUTCOMES:
Change in left ventricular outflow tract velocity time integral | Measured during the basal period and after 1.5 hours of intervention
  Echocardiographic changes in left ventricular outflow tract velocity time integral from the basal period and after 1.5 hours of intervention

SECONDARY OUTCOMES:
Changes in Left Ventricular Ejection Fraction (LVEF) | Measured during the basal period and after 1.5 hours of intervention
  Echocardiographic changes in LVEF from the basal period and after 1.5 hours of intervention
Changes in Global Longitudinal Strain (GLS) | Measured during the basal period and after 1.5 hours of intervention
  Echocardiographic changes in GLS from the basal period and after 1.5 hours of intervention
Changes in S´ Max | Measured during the basal period and after 1.5 hours of intervention
  Echocardiographic changes in S´ Max from the basal period and after 1.5 hours of intervention
Changes in blood pressure | Measured during the basal period and after 1.5 hours of intervention
  Changes in blood pressure from the basal period and after 1.5 hours of intervention
Changes in heart rate | Measured during the basal period and after 1.5 hours of intervention
  Changes in heart rate from the basal period and after 1.5 hours of intervention
Changes in axillary temperature | Measured during the basal period and after 1.5 hours of intervention
  Changes in axillary temperature from the basal period and after 1.5 hours of intervention
Difference in Left Ventricular Ejection Fraction (LVEF) (Healthy vs catabolic conditions) | Measured after 2 hours of basal period
  Echocardiographic difference in LVEF during the basal period between healthy and catabolic conditions (a pooled mean of the two catabolic days, if there is no difference between the first and second time of LPS exposure)
Difference in Global Longitudinal Strain (GLS) (Healthy vs catabolic conditions) | Measured after 2 hours of basal period
  Echocardiographic difference in GLS during the basal period between healthy and catabolic conditions (a pooled mean of the two catabolic days, if there is no difference between the first and second time of LPS exposure)
Difference in S´ Max (Healthy vs catabolic conditions) | Measured after 2 hours of basal period
  Echocardiographic difference in S´ Max during the basal period between healthy and catabolic conditions (a pooled mean of the two catabolic days, if there is no difference between the first and second time of LPS exposure)
Difference in axillary temperature (healthy vs catabolic) | Measured after 2 hours of basal period
  Difference in axillary temperature after 2 hours basal period between healthy and catabolic conditions (a pooled mean of the two catabolic days, if there is no difference between the first and second time of LPS exposure)
Difference in heart rate (healthy vs catabolic) | Measured after 2 hours of basal period
  Difference in heart rate after 2 hours basal period between healthy and catabolic conditions (a pooled mean of the two catabolic days, if there is no difference between the first and second time of LPS exposure)
Difference in blood pressure (healthy vs catabolic) | Measured after 2 hours of basal period
  Difference in blood pressure after 2 hours basal period between healthy and catabolic conditions (a pooled mean of the two catabolic days, if there is no difference between the first and second time of LPS exposure)

CONTACTS AND LOCATIONS:
Overall Officials: Niels Moeller, Professor, Principal Investigator — Aarhus University Hospital and Institute of Clinical Medicine
Locations (1):
- Medical Research Labarotory, DoH, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No